CLINICAL TRIAL: NCT00809861
Title: Volar Locking Plate Versus External Fixator/Cast Fixation for the Treatment of Distal Radius Fractures. A Randomised Controlled Prospective Study
Brief Title: Volar Locking Plate Versus External Fixator/Cast Fixation for the Treatment of Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Base Hospital (Other)
Collaborators: James Cook University, Queensland, Australia (Other)
Responsible Party: Principal Investigator, Dr. Herwig Drobetz, Director Orthopaedics, Mackay Base Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCDRS00407
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): volar locking plating of distal radius fractures
  Interventions: Procedure: volar locking plating
- 2 (Active Comparator)
  Interventions: Procedure: external immobilisation

INTERVENTIONS:
Procedure: volar locking plating — open reduction and internal fixation
  Arms: 1
Procedure: external immobilisation — closed reduction and external fixation
  Arms: 2

SUMMARY:
Aim: Osteosynthesis with locking plate/screws has become increasingly popular in recent years. It is the only treatment option which allows immediate postoperative immobilization. However, compared to conservative treatment or treatment with external fixators, locking plates are very expensive and the operation can be very challenging, even for experienced surgeons. The long-term results of all treatment modalities are equal, which has been shown in numerous studies. However, there are no evidence based studies published yet which look at short-term outcomes. The investigators do feel but do not know that patients who do not need postoperative immobilization return to work significantly earlier or are independent faster than patients whose wrists are immobilized for up to 6 weeks. If that is the case, then the higher costs and risks of the operation are justified, if not, then we have to re-evaluate our indications for using locking distal radius plates distal radius Methods: Group 1: Treatment of distal radius fractures with either volar or dorsal locking plates. No fixation postoperatively, immediate ROM (range of motion) exercises and usage of the wrist in activities of daily life (ADL) allowed.

Radiological and clinical controls 2 weeks, 6 weeks and 12 weeks postoperatively. Endpoints are time to return to work / return to independency (in older people), ROM; Grip strength (with Jamar Dynamometer).

Outcome scores are DASH (Disability of Arm, Shoulder and Hand Score)and PRWE (Patient related wrist evaluation).

Group 2 Treatment of distal radius fractures with either an external fixator +/- K-wires or with K-wires and forearm cast or by cast alone. Main issue is that the wrist is immobilized for a period of 6 weeks. Radiological and clinical controls 2 weeks, 6 weeks and 12 weeks postoperatively. Endpoints are time to return to work / return to independency (in older people), ROM; Grip strength (with Jamar Dynamometer). Outcome scores are DASH and PRWE. Both plating and external fixation / cast fixation are standard and accepted treatment modalities for distal radius fractures. A power analysis indicated that a total sample size of 52 patients randomized equally (1:1) to each treatment arm without any blocking or stratification would provide 80 % statistical power (alpha = .05, beta = .20) to detect a 20% difference in mean DASH and PRWE scores.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fracture
* age > 18

Exclusion Criteria:

* intellectual or mental impairment
* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
20% difference in DASH scores | twelve weeks

SECONDARY OUTCOMES:
return to work | twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Herwig Drobetz, MD, Principal Investigator — Mackay Base Hospital
Locations (1):
- Mackay Base Hospital, Mackay, Queensland, Australia